CLINICAL TRIAL: NCT00165100
Title: Dynamic Area Telethermometry (DAT) as an Auxiliary Imaging Modality in Assessment of Patients With Cancer
Brief Title: Dynamic Area Telethermometry (DAT) as an Imaging Modality in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 99-331
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Malignant Tumors; Subcutaneous Tumors; Lymph Node Tumors
Keywords: DAT; imaging modality
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Procedure: Dynamic Area Telethermometry (DAT)

SUMMARY:
The purpose of this study is to evaluate whether this new method of taking pictures called Dynamic Area Telethermometry (DAT) might be a good way of looking at patients with cancer that is relatively close to the surface of the body.

DETAILED DESCRIPTION:
* The DAT system resembles a video camera which picks up changes in body temperature which may reflect disease-related changes in blood flow to some areas, particularly those involved with tumors.
* Patients with known tumor sites amendable to DAT evaluation will be imaged at the time of staging and at later time points. Thermal profiles will be compared to those of normal adjacent tissues and correlated with the images of the tumors on conventional images.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy
* Primary or secondary tumor location amendable to DAT scanning: subcutaneous tissues
* Older than 15 years of age
* Able to withhold movement for 20 seconds, hold breath for 20 seconds for chest wall lesions and clinically stable acutely

Exclusion Criteria:

* Uncontrolled motion
* Tumors not verified or measurable by standard imaging

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2000-01; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of DAT in tumors detected by conventional imaging and evaluation of therapy induced changes in DAT imaging profile over time.

CONTACTS AND LOCATIONS:
Overall Officials: Milos Janicek, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States